CLINICAL TRIAL: NCT04851886
Title: PostureCheck: A Vision-based Compensatory-posture-detection Tool to Enhance Performance of the BURT Upper-extremity Stroke-therapy
Brief Title: PostureCheck: A Vision-based Compensatory-posture-detection Tool for Robot-assisted Upper-limb Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Barrett Technology (Unknown)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P000197
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either 1) one-on-one robot-assisted upper-limb rehabilitation, and 2) group (up to three subjects per session) robot-assisted upper-limb rehabilitation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Individual robot-assisted upper-limb rehabilitation (Active Comparator): Participants randomized to this arm of the study will undergo 18 sessions of robot-assisted upper-limb rehabilitation. During the sessions, a therapist will administer one-on-one therapy (i.e. each study volunteer will work with a single therapist).
  Interventions: Device: BURT
- Group robot-assisted upper-limb rehabilitation (Experimental): Participants randomized to this arm of the study will also undergo 18 sessions of robot-assisted upper-limb rehabilitation. However, a therapist will administer the intervention as group therapy with up to three subjects participating in the session at the same time. To facilitate the deliver of the therapeutic intervention, the robot will be equipped with a camera system (called PostureCheck) designed to track the quality of the exercises.
  Interventions: Device: BURT + PostureCheck

INTERVENTIONS:
Device: BURT — Robot-assisted upper-limb individual (i.e. one-on-one) rehabilitation will be delivered using the BURT system by Barrett Technology
  Arms: Individual robot-assisted upper-limb rehabilitation
Device: BURT + PostureCheck — Robot-assisted upper-limb group (i.e. up to three subjects) rehabilitation will be delivered using the BURT system by Barrett Technology + PostureChek (a camera-based system to track the quality of the exercises)
  Arms: Group robot-assisted upper-limb rehabilitation

SUMMARY:
The overall objective of this study is to assess whether robot-assisted upper-limb group rehabilitation can be effectively delivered by using a camera-based system equipped with machine learning algorithms to track the quality of the exercise performance and provide feedback accordingly. To address this question, we plan to carry out a randomized clinical trial to compare outcomes in subjects receiving robot-assisted upper-limb rehabilitation during individual (i.e., one-on-one) sessions and in subjects receiving robot-assisted upper-limb rehabilitation during group (i.e., up to three subjects) sessions.

DETAILED DESCRIPTION:
The proposed study is a single-blinded randomized clinical trial to evaluate the effect of using the PostureCheck (a camera-based system equipped with machine learning algorithms to track the quality of the exercise performance) on motor gains in group and individual robot-assisted upper-limb. Study participants (stroke survivors) will be recruited at the Spaulding Rehabilitation Hospital - Boston. Subjects will be randomly assigned to one of the two different groups: individual- or group-therapy using a covariate-adaptive allocation procedure to ensure important covariates, such as baseline Fugl-Meyer Assessment of the Upper Extremity (FMA-UE) scores and proprioceptive deficits, are balanced between groups.

ELIGIBILITY:
Inclusion Criteria:

* Have had a history of ischemic cerebrovascular accident (CVA) within middle cerebral artery (MCA) or anterior cerebral artery (ACA) territory
* CVA occurred between six months and six years ago
* Moderate to severe UE impairment, FMA-UE score between 15 and 45
* Mini-Mental State Examination (MMSE) score >23 and being able to safely follow three-step commands

Exclusion Criteria:

* Advanced musculoskeletal pathology or recent fractures in the impaired UE
* Previous diagnosis of neurological diseases other than stroke
* Severe limitation of passive range of motion or spasticity (Modified Ashworth Scale for spasticity at <3 for UE muscles)
* Hemorrhagic CVA or involvement of the posterior cerebral artery
* Aphasia sufficient to limit ability to express needs or discomfort verbally or non-verbally
* Impaired visual acuity (Severe visual impairments as assessed by the NIH Stroke Scale Visual Field subscale. (score >0))
* Severe hemispatial neglect as assessed by the Line Bisection Test (score >2)
* Severely impaired trunk control (<4)
* Individuals who present with the following on the intended limb:
* Open wounds
* Fragile skin
* Under contact precautions due to an active infection
* Participation in another therapy focused on recovery of the impaired arm
* Subjects with cardiac pacemakers, electronic pumps or any other implanted medical devices, that are not US-certified
* Any Condition that would prevent safe use of the Burt system; such as proprioceptive deficits that impair the ability to process haptic or visual feedback, or unstable shoulder joint as assessed by physical examination
* Current pregnancy (self-report)
* The concern is strictly towards women who are in the 2nd or 3rd trimester and the eventuality of the arm of the BURT accidentally impacting the woman's belly. The system does have safety features (including a virtual safety wall, to keep the device away from the patient's body) but we are taking this as an extra precaution against any potential harm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Fugl-Meyer Assessment - Upper Extremity (FMA-UE) at 7-8 weeks | Data will be collected at baseline and at 7-8 weeks
  Standard assessment of the severity of upper-limb motor impairments

SECONDARY OUTCOMES:
Change from baseline Wolf Motor Function Test (WMFT) at 7-8 weeks | Data will be collected at baseline and at 7-8 weeks
  Standard assessment of functional limitations
Change from baseline Motor Activity Log (MAL) at 7-8 weeks | Data will be collected at baseline and at 7-8 weeks
  Self-report of amount and quality of use of the stroke-affected upper limb

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)

IPD SHARING:
Plan to Share IPD: No